CLINICAL TRIAL: NCT00152035
Title: A Phase III, Multi-center, 12-month, Open-label Safety Study of SPD465 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD).
Brief Title: Safety of SPD465 in Treating Adults With ADHD.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD465-304
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine; Fumigant 93

INTERVENTIONS:
Drug: Neutral salts of dextroamphetamine sulfate, USP, amphetamine sulfate, USP, d-amphetamine saccharate, d, l-amphetamine aspartate monohydrate.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of SPD465 in the treatment of ADHD. The study will also look at how SPD465 affects sleep.

ELIGIBILITY:
Inclusion Criteria:

* Subject satisfied all entry criteria for the antecedent protocol (SPD465-301 or SPD465-303) and completed a minimum of 4 of the 7 weeks of double-blind treatment without experiencing any clinically significant adverse events.
* Subject must be male or non-pregnant female who agrees to comply with using acceptable contraceptive methods.

Exclusion Criteria:

* Subject was terminated from antecedent protocol (SPD465-301 or SPD465-303) for non-compliance and/or experienced a serious adverse event or adverse event resulting in termination from the protocol.
* Comorbid psychiatric diagnosis with significant symptoms such as Axis II disorders or severe Asix I disorders.
* History of seizure, tic disorder, or a current diagnosis and/or family history of Tourette's Disorder.
* Females who are pregnant of lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 505 (Actual)
Dates: Start 2005-03-10 (Actual); Primary Completion 2006-11-07 (Actual); Study Completion 2006-11-07 (Actual)

PRIMARY OUTCOMES:
The evaluation of safety will be based on the occurrence of treatment emergent AEs and specific evaluation of vitals signs, ECG, laboratory and physical examination. | Throughout the study period of approximately 20 months

SECONDARY OUTCOMES:
ADHD-rating scale (ADHD-RS-IV) taken at the Visit 1 and all visits thereafter. | Baseline, Weekly for 4 weeks, and then Monthly for 5 months.
Clinical Global Impression of Improvement scale assessed at Visits 1 through 15/Early Termination (ET). | Baseline, Weekly for 4 weeks, and then Monthly for 5 months.
Pittsburgh Sleep Quality Index (PSQI) - assessed at Visits 1 through 15/ET. | Baseline, Weekly for 4 weeks, and then Monthly for 5 months.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda